CLINICAL TRIAL: NCT05545332
Title: Prospective Multidisciplinary Post-COVID-19 Registry Tyrol
Acronym: PRECISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1450/2021_V2_10_02_2022
Record Dates: First submitted 2022-08-19; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Post COVID-19 Condition
Keywords: post COVID-19 syndrom; long COVID; long term sequelae
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Longitudinal, prospective observational cohort study enrolling patients with persisting symptoms (> 12 weeks) after COVID-19 in a multidisciplinary care model.

DETAILED DESCRIPTION:
Post-COVID-19 syndrome comprises a set of persistent physical, cognitive and/or psychological symptoms that continue for more than 12 weeks after illness and are not attributable to alternative diagnoses. As these symptoms may manifest in all COVID-19 severity grades, even in patients with mild or moderate disease, there is an urgent need for resource allocation in the health care system and accompanied research proposals to understand disease phenotypes and clinical trajectories.

With this prospective multidisciplinary registry, the investigators aim to establish a clinical and researchbased system by providing optimized medical diagnostic and therapeutic approaches in a model region in Austria (Tyrol).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with persistent post COVID symptoms ≥ 12 weeks
* post COVID functional status scale (PCFS) ≥ 2

Exclusion Criteria:

* observation time after infection < 12 weeks
* PCFS < 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be screened by primary physicians in Tyrol (Wester Austria) using the post-COVID-19 functional status (PCFS) scale to assess the functional status, and a symptom checklist for the presence and severity of the 10 most common symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence rates of post-COVID patients requiring multidisciplinary care. | 2 years
  To quantify disease burden by prevalence rates of post-COVID patients requiring multidisciplinary care.
Characterisation of symptom patterns associated with impaired functional status. | up to 24 months
  Characterisation of symptom patterns associated with impaired post covid-19 functional status scale ≥ 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Yes
We provide all of the individual participant data collected during the trial after deidentification and to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning three months after publication and ending five years following article publication.
Access Criteria: Access to researchers who provide a methodologically sound proposal.